CLINICAL TRIAL: NCT04551690
Title: Analysis of Prevalence, Pregnancy Outcomes and Sociodemographic Conditions in Women at Labour With and Without Coronavirus 19 Disease COVID-19 in a Public Hospital in Chile
Brief Title: Prevalence of COVID-19 (Coronavirus Disease 19) in Pregnant Women on Labor in a Public Hospital in Chile (COroNavirus diSease Covid-19 pandEmic iN ChilE)
Acronym: CONSCIENCE
Status: Completed | Type: Observational
Sponsor: Hospital San Juan de Dios, Santiago (Other)
Responsible Party: Principal Investigator, Helga Vera, Principal investigator: Helga Vera von Bargen, Hospital San Juan de Dios, Santiago
Other Study IDs: COVID 19 Pregnancy HSJD Chile
Record Dates: First submitted 2020-07-28; First posted 2020-09-16 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Pregnancy; Covid19; Labor (Obstetrics)--Complications; Demography
Keywords: Pregnancy; Labor; COVID-19; SARS-Cov2; sociodemographic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aim is to assess the prevalence of SARS-COV-2 in unselected pregnant women on labour (or a predictable delivery during next 24 hours), their outcome and sociodemographic conditions.

DETAILED DESCRIPTION:
This is a cross sectional study conducted in Hospital San Juan de Dios, Santiago of Chile. This Hospital attends nearly 4500 births every year. When the COVID-19 pandemia came to Chile, there was no possibility to assess the seroconversion for SARS-Cov2. Currently, it remains unclear the seroprevalence of SARS-Cov-2 in pregnant near to delivery in our country, also its correlation with clinical, perinatal outcomes and sociodemographic characteristics. The project will evaluate these features, collecting nasopharyngeal swab serology in a systematic manner in unselected pregnant women on labor (or a predictable delivery during next 24 hours). Maternal information including clinical data, obstetric history, comorbidities and sociodemographic characteristics acquired from medical records will be correlated to the seroconversion.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women on labor or preterm labor.
* Pregnant women who underwent programmed or emergence cesarean

Exclusion Criteria:

* Stillbirth
* Refusal to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women on labor or preterm labor or who will require interruption of their preg-nancy during the next 24 hours in the Hospital San Juan de Dios in Santiago de Chile between 15 April 2020 and 15 July 2020.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of SARS-CoV-2 in pregnant patients on labor | Through study completion, an average of 4 months
  Determine the prevalence of SARS-CoV-2 in pregnant patients on labor (or a predictable delivery during next 24 hours) with PCR form oropharyngeal swab.
Characterization of clinical features of patients who tested positive for COVID 19. | Through study completion, an average of 4 months
  A questionaire was elaborated to quote all of the following symptoms and were checked at the moment of labour by the residents at charge. The questionaire include following symptoms : presence of fever, cough, dyspnea , headache, myalgia, rhinorrhea, odynophagia and anosmia.
Characterization of living conditions of pregnant women with COVID 19 | Through study completion, an average of 4 months
  Number of bedrooms and number of persons that sleep in that bedroom.

SECONDARY OUTCOMES:
Neonatal hospitalization | Through study completion, an average of 4 months
  Number of days requiring hospitalization in the neonatal unit.
Neonatal weight | Through study completion, an average of 4 months
  Evaluate the neonatal outcome classifying the newborn in adequate for the gestational age, large for gestational age or growth restriction for Parkin. Birth weigt is in grams. We use the Neonatal Growth Charts from Chile.
Perinatal outcomes | Through study completion, an average of 4 months
  Describe the perinatal outcomes of the newborn specifying the Apgar score at delivery.Apgar scores goes form 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Helga Vera von Bargen, physician, Study Chair — Hospital San Juan de Dios AND Universidad de Chile
Locations (1):
- Hospital San Juan de Dios, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- Available data/document: Growth charts of newborns in Chile: helgaisabelv@gmail.com — https://scielo.conicyt.cl/pdf/rcp/v79n4/art03.pdf — helgaisabelv@gmail.com Rev Chil Pediatr 2008; 79 (4): 364-372